CLINICAL TRIAL: NCT05653466
Title: Integrating Complementary Learning Principles in Aphasia Rehabilitation Via Adaptive Modeling (Sub-study 2: Adaptive Trial Scheduling)
Brief Title: Adaptive Trial Scheduling in Naming Treatment for Aphasia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Massachusetts, Amherst (Other); National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, William Evans, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY21120130 (Study 2); 1R01DC019325-01A1 (NIH)
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants responsible for coding data will be masked to treatment condition.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Adaptive spacing, then high-item non-adaptive spacing, then low-item non-adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition
- Adaptive spacing, then low-item non-adaptive spacing, then high-item non-adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition
- High-item non-adaptive spacing, then adaptive spacing, then low-item non-adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition
- High-item non-adaptive spacing, then low-item non-adaptive spacing, then adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition
- Low-item non-adaptive spacing, then high-item non-adaptive spacing, then adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition
- Low-item non-adaptive spacing, then adaptive spacing, then high-item non-adaptive spacing (Experimental): All participants will receive all three naming treatment conditions in a randomized order - this is one possible ordering of those conditions.
  Interventions: Behavioral: Adaptive Spacing Condition; Behavioral: High-Item Non-Adaptive Spacing Condition; Behavioral: Low-Item Non-Adaptive Spacing Condition

INTERVENTIONS:
Behavioral: Adaptive Spacing Condition — Each of the 200 target words for practice are presented on a schedule determined by an algorithm that relies on the pattern of correct vs. incorrect responses for each item. Items in the "active learning" state need to be answered correctly a certain number of times before being categorized as "learned." Each item must be answered correctly 3 times in a row (immediately, then at one-minute and five-minute intervals) before it is categorized as "learned." Then, it will be scheduled at ever-increasing intervals, until answered incorrectly, at which point the item would be returned to the "active learning" state, requiring three correct responses in a row to return again to the "learned" expanding interval state.
Behavioral: High-Item Non-Adaptive Spacing Condition — Each of the 200 target words for practice are presented in sequential order randomized within blocks, with each word presented once before the list repeats.
Behavioral: Low-Item Non-Adaptive Spacing Condition — Each of the 40 target words for practice are presented in sequential order randomized within blocks, with each word presented once before the list repeats.

SUMMARY:
Aphasia is a language disorder caused by stroke and other acquired brain injuries that affects over two million people in the United States and which interferes with life participation and quality of life. Anomia (i.e., word- finding difficulty) is a primary frustration for people with aphasia. Picture-based naming treatments for anomia are widely used in aphasia rehabilitation, but current treatment approaches do not address the long-term retention of naming abilities and do not focus on using these naming abilities in daily life. The current research aims to evaluate novel anomia treatment approaches to improve long-term retention and generalization to everyday life.

This study is one of two that are part of a larger grant. This record is for sub-study 2, which will evaluate the benefits of adaptive trial spacing.

DETAILED DESCRIPTION:
Study 2: Evaluate the benefits of adaptive trial scheduling.

Study design: Investigators will enroll 32 people with aphasia in a randomized within-subjects crossover design comparing an adaptive scheduling condition to two non-adaptive conditions. For each condition, all treatment procedures will be matched except for the number of treated words and the trial spacing manipulation. Participants will receive 10 weeks of computer-based training per condition, with probes administered at baseline and at 1 week, 3 months, and 6 months post-treatment. Condition order will be randomly assigned and counter-balanced across participants. In total, Study 2 will include typically 3-4 (but up to 6) assessment sessions, 120 one-on-one treatment sessions, and 24 baseline and follow-up probe sessions per participant over an ~1-year period, or up to 18 months. All assessment, treatment, and probe sessions will take place via telehealth.

Treatment description: For each condition, all treatment procedures will be matched except for the number of treated words and the trial spacing manipulation. The treatment phase for each of the three conditions will consist of ten weeks of one-on-one treatment four times per week in which the treating clinician will work alongside participants to complete flashcard practice four days a week. The treatment sessions will each last 30 minutes to approximate realistic treatment dosage in outpatient or home health practice settings. Treatment will consist of effortful retrieval practice: on each trial, participants will see a picture of the target and attempt to name it, then rate their naming accuracy by button press. The experimenter will code their response time and perceived accuracy. Finally, the experimenter will code their accuracy which will reveal the target in verbal and written form. If they are unable to name the word correctly, they will be able to replay the answer and repeat it three times prior to moving on to the next trial, per Conroy et al.

ELIGIBILITY:
Inclusion Criteria:

* Existing diagnosis of chronic (>6 months) aphasia subsequent to left hemisphere stroke.
* Impaired performance on 2/8 sections of the Comprehensive Aphasia Test.
* Must have access to a high-speed internet connection and be able to participate in telehealth.

Exclusion Criteria:

* History of other acquired or progressive neurological disease.
* Significant language comprehension impairments
* Unmanaged drug / alcohol dependence.
* Severe diagnosed mood or behavioral disorders that require specialize mental health interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in correct responses in Confrontation Naming of Treated and Untreated Pictured Objects | Initial assessment (pre-treatment), 3 months post-treatment
  Confrontation naming accuracy pictures targeted for each training condition and corresponding untreated items will serve as a primary outcome. Individualized lists for each participant will be selected from a corpus of pictured objects. Performance will be evaluated twice at each timepoint. Change in performance from initial assessment to the 3-month follow-up timepoint on the treated and untreated items will serve as the primary outcome measure.
Change in correct responses in Context Generalization of Treated and Untreated Pictured Objects | Initial assessment (pre-treatment), 3 months post-treatment
  Production of trained words on the context generalization complex scene description task for each training condition and corresponding untreated items will serve as a primary outcome. Words from complex scenes and wordless picture books will be chosen for each participant. These words will consist of a subset of those selected for confrontation naming. Performance will be evaluated twice at each timepoint. Change in performance from initial assessment to the 3-month follow-up timepoint on the treated and untreated items will serve as the primary outcome measure.

SECONDARY OUTCOMES:
Change in core lexicon analysis on the Aphasia Bank Discourse Protocol | Initial assessment (pre-treatment), 3 months post-treatment
  The Aphasia Bank Discourse Protocol is a brief, but thorough set of language tasks which will characterize participants' language at the discourse level. The protocol requires participants to generate discourse samples within the contexts of free speech, a picture description, a story narrative, and procedural discourse. Change in performance in core lexicon analysis on discourse samples from initial assessment to each post-treatment follow up timepoint will serve as a secondary outcome measure.
Change in mean scores on the Aphasia Communication Outcome Measure Short-Form | Initial assessment (pre-treatment), 1 week post-treatment.
  The Aphasia Communication Outcome Measure (ACOM) is a measure of patient-reported "communication functioning," defined as the ability to effectively convey and receive personally relevant messages in natural environments. Results are provided in T scores (sample mean of 50 with a standard deviations of 10), with higher scores indicating better communication functioning.
Score on the Adapted Intrinsic Motivation Inventory for Aphasia | 1 week post-treatment
  The adapted intrinsic motivation Inventory for aphasia is a brief instrument comprised of 7 subscales with a total of 45 items intended to characterize intrinsic motivation in people with aphasia. Each item is scored on a scale of 1-7. Higher total score is associated with higher intrinsic motivation.

CONTACTS AND LOCATIONS:
Overall Officials: William Evans, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- Language Rehab and Cognition Lab, Department of Communication Sciences and Disorders, School of Health and Rehabilitation Sciences, University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing plan for this study includes the publication of discourse measures and other study data on Aphasia Bank (R01-DC008524), a large online repository of aphasia behavioral data that supports a great deal of productive aphasia corpora research. De-identified test scores, treatment, and probe data, and audio and/or video recordings of norming, probe, assessment, and treatment data will be shared to this repository for all study participants.
  Investigators will also make our experimental task files, protocols, and de-identified study data available through Open Science Framework (https://osf.io/) to encourage the replication, collaboration, and expansion of our work by other research groups.
  Last, investigators plan to publish a modeling and statistical package in open-access software, R, which will include functionality for calculating speed-accuracy tradeoff optimality using our multinomial ex-Gaussian response time model approach.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be shared at the time of study publication without planned end to access.
Access Criteria: Anyone who wishes to access the data.